CLINICAL TRIAL: NCT06177938
Title: Lactobreath: A Pilot Study to Diagnose Lactose Intolerance Based on the Exhaled Breath Metabolome
Brief Title: Lactobreath: A Study to Diagnose Lactose Intolerance Using Breath Markers
Acronym: Lactobreath
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ETH Zurich (Other)
Collaborators: Agroscope Liebefeld-Posieux Research Station ALP (Other); Swiss Allergy Centre (Unknown); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NEX_Lactobreath
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-02

CONDITIONS: Lactose Intolerance
Keywords: Lactose; Food Biomarker; Metabolome; Food Intolerance; Microbiota; Breath
MeSH Terms: conditions — Lactose Intolerance; Food Intolerance

STUDY DESIGN:
Intervention Model Description: The study intervention is a single acute postprandial carbohydrate challenge (lactose or glucose) test. Baseline assessments of fecal microbiota composition and usual diet are made on 3 days, within four weeks of the intervention day. Dietary restrictions apply 3 days before the carbohydrate challenge, and participants fast on the morning of the intervention day. The intervention day begins with the collection of baseline urine and breath. Participants are assigned to one of the two carbohydrate challenges. The intervention begins with the ingestion of the carbohydrate solution (25 g of lactose or 13 g glucose) dissolved in 150 mL water, followed by the ingestion of a commercially available gas-sensing capsule to measure intestinal gases. Postprandial breath sampling is conducted over 6 hours for H2 and metabolome analyses. Lactose intolerance symptoms are assessed, and two pools of urine are collected. Intestinal excretion of the gas-sensing capsule marks the end of the intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: NA- No other parties masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactose solution (Experimental): Single ingestion of a lactose solution (25 g lactose dissolved in 150 mL water).
  Interventions: Dietary Supplement: Lactose solution/Glucose solution
- Glucose solution (Placebo Comparator): Single ingestion of a glucose solution (13 g glucose dissolved in 150 mL water).
  Interventions: Dietary Supplement: Lactose solution/Glucose solution

INTERVENTIONS:
Dietary Supplement: Lactose solution/Glucose solution — Single ingestion of a lactose/glucose solution.

SUMMARY:
Food intolerances affect many people and can cause discomfort and dietary challenges. One common cause is difficulty digesting certain carbohydrates called FODMAPs. Diagnosing food intolerance is often done by excluding and then slowly reintroducing these carbohydrates or using a hydrogen breath test, but these methods have limitations.

To address these issues, this project uses the breath we exhale to find markers for lactose intolerance as a model for food intolerance diagnosis. Our aim is to identify breath markers for lactose tolerance and intolerance and link them to metabolic traits, including those found in urine. We use a real-time breath analysis method and a special sensor to measure gases in the digestive system, and we also explore genetic factors using saliva samples.

This project aims to help clinicians better identify patients who should follow low FODMAP diets and provide non-invasive breath tests to predict how patients will respond to these diets. It will also advance the use of breath analysis for personalized nutrition, contributes to the broader field of food intolerance research, and has the potential to benefit millions of individuals worldwide.

DETAILED DESCRIPTION:
Genetic and lactose tolerance screening For all eligible participants, a screening home test will be conducted. The home screening test kit will contain lactose powder and accompanying information in order for the subjects to conduct a lactose tolerance test (according to the LHBT protocol) at home. The test will be adapted from recent guidelines (https://www.esnm.eu/guidelines.html) that propose the use of 25g of lactose for lactose tolerance testing, including a questionnaire to quantitatively assess symptoms. The home screening test kit will also provide material to collect a saliva sample to determine genetic polymorphisms commonly modulating LP.

A total of 120 participants will be selected and distributed into three groups based on their LP genetic profiles and response to the ingestion of 25 g of lactose (lactose solution):

* 24 genetically LP subjects with no GI symptoms in response to the ingestion of lactose (group 1)
* 24 genetically lactase-non-persistent (LNP) subjects with no GI symptoms in response to the ingestion of lactose (group 2)
* 72 genetically LNP subjects with any GI symptoms in response to lactose ingestion (group 3).

Study procedures Baseline measures: For each subject, baseline measurement of microbiota and diet will be made within four weeks of the intervention day. The assessment of diet and the genomic characterization of the fecal microbiota will be performed in parallel with repeated measures

* Four 24 h dietary recalls will be completed using an adapted version of the myfood24 online platform on four consecutive days, during days -30 to -7, before the intervention day
* Three fecal samples will be collected by the participants at home, ideally on three consecutive days, on days +1, +2, and +3 relative to the first 24 h dietary recall.

Intervention day: The diet of all selected participants will be restricted for the three days before the carbohydrate challenge test day to ensure that all FODMAPs are avoided with a standardized diet provided to the participants for the three days before the test.

On the morning of the test day, the participants will be asked to collect their first test sample, the morning urine and consume 300 mL of water at home. Upon arrival in the test laboratory, the participants will deliver a further urine sample and baseline breath samples for the breath metabolome and hydrogen breath test. The urine samples will be used for metabolomics analysis and, in the case of female participants, for a pregnancy test. Participants with a positive pregnancy test will be excluded.

The participants will also fill out the questionnaire on LI (as used for the screening survey) to describe symptoms of LI before the test (baseline symptoms).

The 120 participants will be assigned to one of the two carbohydrate challenges using stratified randomization based on the three groups defined by the pre-screening tests. 100 participants will be assigned to the experimental intervention (lactose). The remaining 20 participants (4 participants from each groups 1 and 2 and 12 participants from group 3) will be assigned to the control intervention (glucose). The participants and investigators will be blinded during testing to the type of carbohydrate solution assigned.

For each participant, the carbohydrate solution will need to be consumed in a time-lapse of 5 min. Following the solution intake, participants will be asked to rinse their mouths with a standard quantity of water (500 mL) to avoid the detection of solution-relevant residual molecules in the oral cavity. The participants will swallow a commercially available gas-sensing capsule within the 5 minutes following the lactose or glucose solution intake to monitor intestinal gases and GI transit time.

Postprandial breath, exhaled breath condensate (EBC) and urine samples will then be collected at predefined times during the 6 h following consumption of the assigned test product. Breath sampling will be performed using a secondary electrospray ionization source coupled to a high-resolution mass spectrometry system (SESI-HR-MS) for direct and real-time detection of volatile organic compounds (VOC) and using an H2 breath sensor (e.g. QuinTron BreathTracker Digital Microlyzer) for detection of exhaled hydrogen. EBC samples will be collected using a spirometry filter connected to a glass cold trap cooled to -78°C. In addition, the participants will fill out the questionnaire for symptoms of LI to describe the symptoms during the 6 h postprandial assessment .

To normalize participants' hydration, particularly to facilitate the urine collection, the participants will be offered a standardized quantity of water based on their body weight to be consumed in regular portions during the post-ingestion period. No other foods or fluids will be permitted during the laboratory testing.

Intestinal excretion of the gas-sensing capsule will mark the end of the intervention. A follow-up visit to confirm the excretion of the gas-sensing capsule will conclude the study.

Additional subjects will be recruited should the number of participants completing the lactose and glucose tests fall below the targeted numbers.

ELIGIBILITY:
Inclusion criteria:

* Men and women
* Swiss and non-Swiss living in the Zurich area (if necessary, beyond Zürich in Switzerland),
* Ability/desire to provide informed consent and partake in the procedures of the study
* Aged 18-65 years at screening
* Agreement to refrain from all other treatments and products used for dairy intolerance (e.g., Lactaid® dietary supplements) during study involvement
* Willing to return for all study visits and complete all study-related procedures, including fasting before and during the intervention
* Able to understand and provide written informed consent in English and/or German.

Exclusion criteria:

* Allergic to milk
* Currently pregnant
* Currently lactating
* Cigarette smoking or other use of tobacco or nicotine-containing products within 3 months of screening
* Diagnosed with any of the following disorders known to be associated with abnormal GI motility: gastroparesis, amyloidosis, neuromuscular diseases (including Parkinson's disease), collagen vascular diseases, alcoholism, uremia, malnutrition, or untreated hypothyroidism
* History of surgery that alters normal GI tract function, including but not limited to: GI bypass surgery, bariatric surgery, gastric banding, vagotomy, fundoplication, pyloroplasty (N.B. history of uncomplicated abdominal or GI surgeries such as removal of an appendix >12 months before screening will not be excluded)
* Suspected obscure GI bleeding
* Past or present: organ transplant, chronic pancreatitis, pancreatic insufficiency, symptomatic biliary disease, coeliac disease, diverticular disease, inflammatory bowel disease, strictures (suspected or known), fistulas, or any GI obstruction, gastroparesis, history of gastric bezoar or any other medical condition with symptoms that could confound collection of adverse events
* Diabetes mellitus
* Congestive heart failure
* Human immunodeficiency virus, hepatitis B, or hepatitis C
* Body mass index > 35 kg/m2
* Swallowing disorders or dysphagia to food or pills
* Presence of implantable or portable electro-mechanical medical devices (e.g. pacemakers)
* Recent bowel preparation for endoscopic or radiologic investigation within 4 weeks of screening (e.g., colonoscopy preparation)
* Chronic antacid and/or proton pump inhibitor use
* Recent use of systemic antibiotics, defined as use within 2 months prior to screening
* History of ethanol (alcohol) and/or drug abuse in the past 12 months
* Patients with severe irritable bowel syndrome (IBS) (i.e., IBS Symptom Severity Score >400)
* Dietary restrictions including vegan or vegetarian diet.
* Any other conditions/issues noted by the study staff and/or Principal Investigator that would impact participation and/or protocol compliance.
* Previous enrollment in another clinical trial within the last 3 months.
* Results of the screening test showing GI symptoms in response to lactose ingestion and genetic LP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of the breath profile associated with lactose malabsorption (lactobreath profile) | Breath samples will be collected at 9 time points following the ingestion of lactose (15 min, 30 min, 60 min, 90 min, 120 min, 180 min, 240 min, 300 min, and 360 min).
  Selected metabolites identified from exhaled breath after lactose intake that can collectively discriminate clinical traits associated with lactose malabsorption. Several parameters with be assessed: sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), the likelihood ratio of a positive test (LR+), the likelihood ratio of a negative test (LR-).

SECONDARY OUTCOMES:
Urine metabolome | Two pooled postprandial timepoints following lactose intake (0-3h and 3-6h)
  Metabolites identified in urine samples using GC-qTOF (including lactose and its metabolites, galactose, galactitol, and galactonate).
Metabolome of exhaled breath condensate (EBC) samples | 9 postprandial timepoints following lactose intake (15 min, 30 min, 60 min, 90 min, 120 min, 180 min, 240 min, 300 min, and 360 min)
  Metabolites identified in EBC samples using standardized LC-MS methods (reversed-phase and HILIC) and GC-MS.
Hydrogen breath test | 9 postprandial timepoints following lactose intake (15 min, 30 min, 60 min, 90 min, 120 min, 180 min, 240 min, 300 min, and 360 min)
  Dynamic assessment of the hydrogen in breath after dietary exposure using hydrogen breath sensor
Intestinal gases and GI transit assessment | Semi-continuous (every 20 seconds) postprandial assessment following lactose intake until excretion of the capsule
  Dynamic assessment of the environment of the intestine via a commercial gas-sensing capsule to evaluate intestinal gas concentrations (H2, O2, CO2, and CH4), pH and GI transit.
Clinical symptoms of lactose intolerance | 5 postprandial timepoints following lactose intake (30 min, 60 min, 120 min, 180 min, and 360 min)
  Standardized questionnaire previously validated for the target population

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All results from the study will be published publicly and accessible without restrictions, in accordance with the SNSF open access policy. The accepted version will be deposited in the ETH Research Collection (www.research-collection.ethz.ch), the so-called "green way" for open access. The microbiota data will be published at the European Nucleotide Archive (https://www.ebi.ac.uk/ena/browser/home) after all relevant data have been published. Details of the study design will be available through the phenotype database. All other data will be accessible from within our organization, ETH Zurich. If an external scientist wishes to access the data, there are straightforward options to do so (for example, setting up a guest account at ETH that allows access via a VPN account). Such access will be granted upon reasonable request.

REFERENCES:
- [Derived] Giannoukos S, Burton-Pimentel KJ, Guillod R, Vergeres G, Pohl D. Exploring exhaled breath biomarkers for lactose intolerance diagnosis: the Lactobreath pilot study protocol. BMJ Open. 2025 Aug 3;15(8):e107256. doi: 10.1136/bmjopen-2025-107256. PMID 40754327